CLINICAL TRIAL: NCT05720897
Title: Comparing Brief Relaxation Period to Virtual Reality Period in Reducing Dental Anxiety Prior to Root Canal Treatment; a Randomized Control Trial
Brief Title: Comparing Brief Relaxation Period to Virtual Reality Period in Reducing Dental Anxiety Prior to Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Stuart Schrader, Clinical Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 17053
Record Dates: First submitted 2023-01-09; First posted 2023-02-09 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Auditory Alone Brief Relaxation (Experimental): Participants randomized to this arm will receive earphones to listen to a guided brief relaxation recording, focusing on breathing and a body scan, prior to their dental procedure.
  Interventions: Other: Auditory Alone
- Relaxation Virtual Reality (Experimental): Participants will receive virtual reality goggles and choose a scene of their liking to experience, prior to their dental procedure.
  Interventions: Device: Relaxation Virtual Reality

INTERVENTIONS:
Other: Auditory Alone — Participants randomized to this arm will receive earphones to listen to an 8 minute guided brief relaxation recording, focusing on breathing and a body scan. Participants will listen to the recording prior to their dental procedure.
  Other Names: ABR
  Arms: Auditory Alone Brief Relaxation
Device: Relaxation Virtual Reality — Participants randomized to this arm will receive will receive virtual reality goggles and choose a scene of their liking to experience. Participants will choose from 11 different themed environments (such as savannah, beach, meadow, or space), and will experience the chosen virtual reality environment for 8 minutes. Participants will complete the virtual reality intervention prior to their dental procedure.
  Other Names: RVR
  Arms: Relaxation Virtual Reality

SUMMARY:
The goal of this study is to evaluate non-drug approaches to reducing dental anxiety prior to non-surgical root canal treatment. This will be done by comparing two relaxation methods which will be performed immediately prior to scheduled, clinical non-surgical root canal treatment. Measures of anxiety will be evaluated prior to, and after, the relaxation intervention, as well as after the non-surgical root canal treatment is completed. Participation in the study is completed in a single study visit.

DETAILED DESCRIPTION:
Fifty-eight participants who needed non-surgical root canal treatment were randomly assigned into 2 groups of ABR and VRR. One group received earphones to listen to a guided brief relaxation recording, focusing on a body scan of tense points with diaphragmatic breathing. The other group received Meta 2 virtual reality headsets to listen and watch a 360 inclusive and integrative experience of ambient music, high resolution graphic illustrations and immersive scenery. Participants self-reported levels of anxiety were assessed prior to and post treatment by conducting evaluations using the State Trait Anxiety Indicator (STAI-State & Trait) and the use of both a self-reported Visual Analog Scale (VAS) as well as by assessing objective secondary biometrics of anxiety of heart rate (HR) and Blood Pressure (BP) pre intervention, post intervention and following treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* requires non-surgical root canal treatment
* is able to independently provide informed consent for root canal treatment
* proficient in English

Exclusion Criteria:

* history of vertigo or severe motion sickness
* history of severe psychiatric disease
* history of seizures, concussions, or severe neurological conditions
* visual or hearing impairments
* cardiac pacemaker or defibrillator
* will require nitrous oxide sedation, nor pharmacologic anxiolytics or sedatives for dental treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Schrader, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, School of Dentistry, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Relaxation Virtual Reality: Participants will receive virtual reality headset and choose a scene of their liking to experience, prior to their dental procedure.
  Relaxation Virtual Reality: Participants randomized to this arm will receive will receive virtual reality headsets and choose a scene of their liking to experience. Participants will choose from 11 different themed environments (such as savannah, beach, meadow, or space), and will experience the chosen virtual reality environment with accompanying music for 8 minutes. Participants will complete the virtual reality intervention prior to their dental procedure.
Period: Overall Study
Arm/Group | Auditory Alone Brief Relaxation | Relaxation Virtual Reality
Started | 30 | 30
Completed | 28 | 30
Not Completed | 2 | 0
Not completed — Two patients did not complete Endodontic Treatment & there was technical VR difficulties for pts. | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auditory Alone Brief Relaxation | Relaxation Virtual Reality | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Customized [Mean (Full Range); unit: Years] | 41.9 [19 to 74] | 45.9 [21 to 81] | 43.9 [19 to 81]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Male, Female and Open Reporting for Additional Identification
  Participants
    Gender Identification: Male | 10 | 16 | 26
    Gender Identification: Female | 18 | 13 | 31
    Gender Identification: Additional Identification | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 23 | 26 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 5 | 13
  White | 16 | 17 | 33
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
STAI-S [Mean (Standard Deviation); unit: units on a scale] — The State Trait Anxiety Inventory State sub-scale (STAI-S) is a 20 item sub-scale questionnaire which measures subjective self-reported feelings of state anxiety. Responses for each item include four possible responses that range from "not at all" to "very much" and which correlate to a numerical value. Scores range from 20 to 80. A score of 45-80 indicates "high anxiety": 38-44 indicate "moderate anxiety": 20-37 indicate low or no anxiety.
  units on a scale | 33.75 (9.87) | 35.13 (10.64) | 34.46 (10.21)
STAI-T [Mean (Standard Deviation); unit: units on a scale] — The State Trait Anxiety Inventory Trait sub-scale (STAI-T) is a 20 item sub-scale questionnaire which measures subjective self-reported feelings of trait anxiety. Responses for each item include four possible responses that range from "not at all" to "very much" and which correlate to a numerical value. Scores range from 20 to 80. A score of 45-80 indicates "high anxiety": 38-44 indicate "moderate anxiety": 20-37 indicate low or no anxiety.
  units on a scale | 31.86 (10.94) | 33.77 (10.22) | 32.85 (10.52)
Visual Analogue Scale (VAS) for Anxiety [Mean (Standard Deviation); unit: units on a scale] — Visual Analogue Scale for Anxiety: 0 Least Anxiety to 10 Most Anxiety
  units on a scale | 2.68 (2.44) | 2.43 (2.05) | 2.55 (2.23)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — CDC Normal Overall Mean Systolic Blood Pressure <120 Elevate risk for hypertension: >129 Stage 1 hypertension: 130-139 Stage 2 hypertension 140-180 Potential hypertensive Crisis: >180
  mmHg | 134.68 (15.63) | 131.90 (16.81) | 133.24 (16.17)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Accord to CDC:
  Normal - <80 At Risk - 80-89 for Hypertension Higher Risk - >90 for Hypertension
  mmHg | 82.36 (10.29) | 81.83 (10.65) | 82.09 (10.39)
Heart Rate [Mean (Standard Deviation); unit: bpm] — According to the CDC
  Avg resting heart rate for adults - 60-100 beats per minute (BPM) Above 100 - may need medical attention Above 140 - may be dangerous
  bpm | 77.82 (11.53) | 76.97 (11.89) | 77.38 (11.62)

OUTCOME MEASURES:

1. Primary Outcome: State-Trait Anxiety Inventory State Sub-scale (STAI-S) Score at the End of the Appointment
Description: STAI-S is a 20 item sub-scale questionnaire which measures subjective self-reported feelings of state anxiety. Responses for each item include four possible responses that range from "very much" to "not at all" and which correlate to a numerical value. Scores range from 20 to 80. A score of 45-80 indicates "high anxiety": 38-44 indicate "moderate anxiety": 20-37 indicate low or no anxiety.
Time Frame: End of the appointment, approximately 90+ minutes after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Auditory Alone Brief Relaxation: Participants randomized to this arm received earphones to listen to a guided brief relaxation recording, focusing on breathing and a body scan, prior to their dental procedure.
  Auditory Alone: Participants randomized to this arm received earphones to listen to an 8 minute guided brief relaxation recording, focusing on breathing and a body scan. Participants listened to the recording prior to their dental procedure.
- Relaxation Virtual Reality: Participants will receive virtual reality headset and choose a scene of their liking to experience, prior to their dental procedure.
  Relaxation Virtual Reality: Participants randomized to this arm will receive will receive virtual reality headset and choose a scene of their liking to experience. Participants choose from 11 different themed environments (such as savannah, beach, meadow, or space), and experienced the chosen virtual reality environment for 8 minutes. Participants completed the virtual reality intervention prior to their dental procedure.
Arm/Group | Auditory Alone Brief Relaxation | Relaxation Virtual Reality
Number analyzed (Participants) | 28 | 30
units on a scale | 27.39 (7.84) | 29.37 (9.0)
Statistical Analysis 1: Comparison: Auditory Alone Brief Relaxation vs Relaxation Virtual Reality; The study has an 80% power to detect changes in patient's self-reported anxiety as measured by their responses to the psychometrically validated STAI-S & T instrument of 3.6 within each group (with an effect size of 0.55) and differences of a 5.0 between groups (with an effect size of 0.77); Test type: Superiority; p = .399, Wilcoxon (Mann-Whitney) — The calculations are based on a Mann Whitney calculation

2. Primary Outcome: Visual Analog Score (VAS) at the End of the Appointment
Description: The VAS will be a single question in which the participant is asked to assign and report a numerical value to the amount of anxiety one is feeling in the moment. It consists of a 10 point scale, with one symbolizing no anxiety and 10 symbolizing unbearable anxiety.
Time Frame: End of the appointment, approximately 90+ minutes after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auditory Alone Brief Relaxation | Relaxation Virtual Reality
Number analyzed (Participants) | 28 | 30
units on a scale | 0.96 (0.96) | 1.17 (1.97)

3. Primary Outcome: Systolic Blood Pressure (SBP) at the End of the Appointment
Description: BP will be measured three times during the single study visit: at enrollment (prior to the assigned relaxation intervention), at the end of the assigned relaxation intervention, and at the end of the appointment.
Time Frame: End of the appointment, approximately 90+ minutes after baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Auditory Alone Brief Relaxation | Relaxation Virtual Reality
Number analyzed (Participants) | 28 | 30
mmHg | 142.64 (20.03) | 137.47 (22.45)

4. Primary Outcome: Diastolic Blood Pressure (DBP) at the End of the Appointment
Description: as for outcome 3
Time Frame: End of the appointment, approximately 90+ minutes after baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Auditory Alone Brief Relaxation | Relaxation Virtual Reality
Number analyzed (Participants) | 28 | 30
mmHg | 90.00 (12.56) | 85.97 (15.48)

5. Primary Outcome: Heart Rate (HR) at the End of the Appointment
Description: HR will be measured three times during the single study visit: at enrollment (prior to the assigned relaxation intervention), at the end of the assigned relaxation intervention, and at the end of the appointment.
Time Frame: End of the appointment, approximately 90+ minutes after baseline
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Auditory Alone Brief Relaxation | Relaxation Virtual Reality
Number analyzed (Participants) | 28 | 30
bpm | 72.89 (9.09) | 72.17 (10.90)

6. Primary Outcome: State-Trait Anxiety Inventory Trait Sub-scale (STAI-T) Score at the End of the Appointment
Description: STAI-T is a 20 item sub-scale questionnaire which measures subjective self-reported feelings of trait anxiety. Responses for each item include four possible responses that range from "not at all" to "very much" and which correlate to a numerical value. Scores range from 20 to 80. A score of 45-80 indicates "high anxiety": 38-44 indicate "moderate anxiety": 20-37 indicate low or no anxiety.
Time Frame: End of the appointment, approximately 90+ minutes after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auditory Alone Brief Relaxation | Relaxation Virtual Reality
Number analyzed (Participants) | 28 | 30
units on a scale | 30.18 (11.55) | 29.90 (8.53)

ADVERSE EVENTS:
Time Frame: The 1 day in which data was collected.
Groups:
- Relaxation Virtual Reality: Participants will receive virtual reality headsets and choose a VR scene of their liking to experience, prior to their dental procedure.
  Relaxation Virtual Reality: Participants randomized to this arm will receive will receive virtual reality headsets and choose a scene of their liking to experience. Participants will choose from 11 different themed environments (such as savannah, beach, meadow, or space), and will experience the chosen virtual reality environment with accompanying music for 8 minutes. Participants will complete the virtual reality intervention prior to their dental procedure.
Arm/Group | Auditory Alone Brief Relaxation | Relaxation Virtual Reality
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05720897/Prot_SAP_000.pdf